CLINICAL TRIAL: NCT01242358
Title: Clinical Value of Advanced Patient Monitoring Using Capnography With Analysis of the Integrated Pulmonary Index During Percutaneous Endoscopic Gastrostomy.
Brief Title: Capnography During Percutaneous Endoscopic Gastrostomy (PEG)
Acronym: PEG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Andrea Riphaus, Clinical value of capnography During Percutaneous Endoscopic Gastrostomy (PEG), Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Capno-PEG 2010
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: In the Study the Value of Capnography for Avoiding Complications During Sedation for PEG is Evaluated.
Keywords: hypoxaemia - capnography - integrated pulmonary index - PEG
MeSH Terms: interventions — Capnography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capnography (Experimental): Arm with capnographic monitoring
  Interventions: Device: Capnography
- Standard monitoring (Placebo Comparator): Standard monitoring
  Interventions: Device: Standard monitoring

INTERVENTIONS:
Device: Capnography — Capnographic monitoring
  Arms: Capnography
Device: Standard monitoring — Standard monitoring
  Arms: Standard monitoring

SUMMARY:
In this randomized controlled trial the utility of capnography gets evaluated. Hypoxemia may occur during sedation with midazolam and propofol. Whether hypoxemia may be prevented by an additional capnographic monitoring is subject of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Scheduled for PEG with propofol sedation

Exclusion Criteria:

* No informed consent
* ASA V
* Emergency endoscopy
* Preexisting hypotension, bradycardia or hypoxemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Hypoxemia | From the beginning to the end of the PEG procedure, i.e. from 0h to approximately 2h

SECONDARY OUTCOMES:
Further complications | From the beginning to the end of the PEG procedure, i.e. from 0h to approximately 2h

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Riphaus, MD, Principal Investigator — Ruhr-Universität Bochum
Locations (3):
- Germany (3):
  - Ruhr Universität Bochum, Bochum
  - Technische Universität München, München
  - Deutsche Klinik für Diagnostik, Wiesbaden

REFERENCES:
- [Result] Vargo JJ, Zuccaro G Jr, Dumot JA, Conwell DL, Morrow JB, Shay SS. Automated graphic assessment of respiratory activity is superior to pulse oximetry and visual assessment for the detection of early respiratory depression during therapeutic upper endoscopy. Gastrointest Endosc. 2002 Jun;55(7):826-31. doi: 10.1067/mge.2002.124208. PMID 12024135